CLINICAL TRIAL: NCT05488678
Title: VNRX-7145-103: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Ceftibuten/VNRX-7145 in Participants With Varying Degrees of Renal Function
Brief Title: Ceftibuten/VNRX-7145 in Participants With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VNRX-7145-103; 272201600029C-P00026-9999-1 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ceftibuten

STUDY DESIGN:
Intervention Model Description: The study will enroll approximately 32 participants assigned to groups based on renal function.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 - Control (Experimental): Healthy control participants will be matched by gender, age, and BMI to participants with renal impairment
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Group 2 - Mild Renal Impairment (Experimental): Mild Renal Impairment
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Group 3 - Moderate Renal Impairment (Experimental): Moderate Renal Impairment
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Group 4 - Severe Renal Impairment (Experimental): Severe Renal Impairment
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Group 5 - End Stage Renal Disease (Experimental): End Stage Renal Disease undergoing chronic intermittent hemodialysis
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten

INTERVENTIONS:
Drug: VNRX-7145 — single oral dose
Drug: Ceftibuten — single oral dose

SUMMARY:
This is an open-label, multicenter, parallel-group study in participants with normal renal function, mild, moderate, or severe renal impairment, or end stage renal disease (ESRD) undergoing standard intermittent dialysis. The pharmacokinetics (PK) of the inactive prodrug VNRX-7145, its active parent drug VNRX-5236, and ceftibuten will be evaluated after a single oral dose of ceftibuten/VNRX-7145.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-82 years
* Males or non-pregnant, non-lactating females
* Body mass index (BMI): ≥18.5 kg/m2 and ≤40.0 kg/m2
* Laboratory values meeting defined entry criteria

Subjects with normal renal function (Group 1) must also meet the following criteria:

• Match to one or more participants with renal impairment by gender, age, and BMI

Subjects with renal impairment (Groups 2-5) must also meet the following criteria:

• Stable, pre-existing renal impairment

Exclusion Criteria:

* History of drug allergy or hypersensitivity to penicillin, cephalosporin, or beta-lactam antibacterial drug
* Congenital or acquired immunodeficiency syndrome
* Major adverse cardiovascular event within one year of dosing
* Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-120 hours post dose
  Maximum plasma concentration, determined directly from individual concentration time data
AUC0-inf | 0-120 hours post dose
  Area under the plasma concentration time curve from time zero extrapolated to infinity based on collected PK
Number of subjects with adverse events | 8 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (3):
- United States (3):
  - Advanced Pharma, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota